CLINICAL TRIAL: NCT00955617
Title: Intra-individual Efficacy Evaluation of DOTAREM®-Enhanced MRA Compared to GADOVIST®-Enhanced MRA in the Diagnosis of Clinically Significant Abdominal or Lower Limb Arterial Diseases
Brief Title: DOTAREM®-Enhanced MRA Compared to GADOVIST®-Enhanced MRA in Patients With Abdominal or Lower Limb Arterial Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: DGD-44-052
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Results first posted 2012-11-02 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Peripheral Arterial Disease
Keywords: Dotarem; Gadovist; Peripheral arterial disease; MRA
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dotarem / Gadovist (Experimental): Contrast-enhanced MRA - Imaging examination contrast enhanced-MRA first with Dotarem in period 1 then with Gadovist in period 2
  Interventions: Other: Contrast-enhanced MRA - Imaging examination
- Gadovist / Dotarem (Experimental): Contrast-enhanced MRA - Imaging examination contrast enhanced-MRA first with Gadovist in period 1 then with Dotarem in period 2
  Interventions: Other: Contrast-enhanced MRA - Imaging examination

INTERVENTIONS:
Other: Contrast-enhanced MRA - Imaging examination — Administration of 0.1 mmol/kg of contrast product (Dotarem and Gadovist)
  Other Names: Dotarem-enhanced MRA; Gadovist-enhanced MRA

SUMMARY:
This study is an intra-individual comparison of DOTAREM®-enhanced MRA and GADOVIST®-enhanced MRA in the diagnosis of clinically significant abdominal or lower limb arterial diseases.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, aged ≥ 18 years
* Patient suffering from Peripheral Arterial Occlusive Disease (PAOD) stage II or III.

Exclusion Criteria:

* Patients with severely impaired renal function with an eGFR (MDRD) < 50ml/min (eGFR based on recent serum creatinine and MDRD formula - younger than 21 days).
* Patient planned to undergo therapeutic intervention in the vessels of interest between the two MRA procedures.
* Patient who had a major cardiovascular event within 30 days prior to the inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guerbet, Study Director — Guerbet
Locations (1):
- Guerbet, Roissy CDG, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Dotarem Then Gadovist: Cross over administration, patient received first Dotarem enhanced-MRA (MRA1) and then Gadovist enhanced-MRA (MRA2)
- Gadovist Then Dotarem: Cross over administration: patient received first Gadovist enhanced-MRA (MRA1) and then Dotarem enhanced-MRA (MRA2)
Period: First MRA (Between Day0 and Day21)
Arm/Group | Dotarem Then Gadovist | Gadovist Then Dotarem
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second MRA (Between Day 1 and Day 51)
Arm/Group | Dotarem Then Gadovist | Gadovist Then Dotarem
Started | 10 | 10
Completed | 7 | 7
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — technical incident | 0 | 1
Not completed — conventional angiography | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All Patients received both product Dotarem and Gadovist during 2 enhanced-MRA. Demographic analysis was performed on the global population.
Arm/Group | All Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 61.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Region of Enrollment [Number; unit: participants]
  Germany | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Image Quality of MRA Images
Description: Number of images quoted with excellent and more than adequate quality in each group.
  Image quality will be assessed on a 5-point scale:
  1. Excellent
  2. More than adequate
  3. Adequate
  4. Less than adequate
  5. Non-diagnostic
  Each image is analysed by 4 readers.
Time Frame: MRA examination
Population: descriptive and pilot study, no number of participants calculation performed
Measure: Number; unit: Images
Units Other Than Participants: cases (4 evaluations per image)
Groups:
- Dotarem: Evaluation performed on Dotarem enhanced MRA images
- Gadovist: Evaluation performed on Gadovist enhanced MRA images
Arm/Group | Dotarem | Gadovist
Number analyzed (Participants) | 14 | 14
Number analyzed (cases (4 evaluations per image)) | 56 | 56
Images | 56 | 48

2. Secondary Outcome: Diagnostic Confidence
Description: Number of High/Excellent diagnostic confidence. Level of diagnostic confidence assessed on a 5-point scale by patient: nil, poor, moderate, high, excellent.
  Each image is analysed by 4 readers.
Time Frame: MRA examination
Population: Descriptive study - No calculation
Measure: Number; unit: Images
Units Other Than Participants: cases (4 evaluations per image)
Arm/Group | Dotarem | Gadovist
Number analyzed (Participants) | 14 | 14
Number analyzed (cases (4 evaluations per image)) | 56 | 56
Images | 55 | 50

3. Secondary Outcome: Signal Intensity
Description: Signal to Noise ratio (SNR): SNR = SIa /NO SIa is the signal intensity measured in the ROI positioned in the artery. NO is noise defined as the standard deviation (SD) of signal intensity measured in the subtraction image (of the two non-enhanced scans) at the same location as the arterial ROI is to be measured.
Time Frame: MRA examination
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Dotarem | Gadovist
Number analyzed (Participants) | 14 | 14
Ratio | 23 (10) | 26 (11)

ADVERSE EVENTS:
Groups:
- Dotarem MRA: Patients who received a Dotarem enhanced-MRA
- Gadovist MRA: Patients who received a Gadovist enhanced-MRA
Arm/Group | Dotarem MRA | Gadovist MRA
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Limitation of the study: descriptive study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less